CLINICAL TRIAL: NCT05756504
Title: "NSAIDs vs. Opiates: Which is More Effective in Managing Pain in Mild to Moderate Acute Pancreatitis? A Randomized Controlled Trial"
Brief Title: "NSAIDs vs. Opiates: Which is More Effective in Managing Pain in Mild to Moderate Acute Pancreatitis?
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hayatabad Medical Complex (Other Government)
Responsible Party: Principal Investigator, Musarrat Hussain, Assistant Professor, Department of Surgery, Hayatabad Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMC-QAD-F-1202
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Ketorolac; Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSAIDs (Experimental): Patients in this arm will be given ketorolac injection 30 mg IV x TDS for pain management of mild to moderate acute pancreatitis
  Interventions: Drug: Ketorolac
- Opioids (Experimental): Patients in this arm will be given injection tramadol IV x TDS for pain management of mild to moderate acute pancreatitis
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Ketorolac — Injection ketorolac 30 mg IV x TDS will be given to each patient in each group.
  Arms: NSAIDs
Drug: Tramadol — Injection Tramadol 25-50 mg IV x TDs wil be given to each patient in this group. Maximum dose will be 400 mg/ day
  Arms: Opioids

SUMMARY:
Acute pancreatitis is a painful and potentially life-threatening condition that affects the pancreas, a glandular organ responsible for producing digestive enzymes and hormones. The condition is typically characterized by sudden inflammation of the pancreas that can cause severe abdominal pain, nausea, and vomiting. Treatment for acute pancreatitis usually involves supportive care, pain management, and sometimes, hospitalization.

Nonsteroidal anti-inflammatory drugs (NSAIDs) and opioids are two of the most commonly used classes of pain medication for the management of acute pancreatitis. While both drugs are effective in reducing pain, they have different mechanisms of action and potential side effects. NSAIDs work by reducing inflammation and pain by inhibiting the activity of cyclooxygenase (COX) enzymes, whereas opioids work by binding to specific receptors in the brain and spinal cord to block the transmission of pain signals.

Despite their widespread use, there is a lack of consensus regarding which medication is more effective for the management of acute pancreatitis, particularly in mild to moderate cases. Some studies have suggested that NSAIDs may be more effective for reducing pain in acute pancreatitis, while others have suggested that opioids may be more effective in providing pain relief. Moreover, there is a concern regarding the potential for adverse events associated with the use of opioids, such as respiratory depression, addiction, and constipation.

Therefore, this study aims to compare the efficacy and safety of NSAIDs and opioids in the management of mild to moderate acute pancreatitis. This will be a randomized clinical trial, which will involve the recruitment of patients with mild to moderate acute pancreatitis who will be randomized to receive either an NSAID or an opioid for pain management. The primary outcome of this study will be the reduction in pain score measured using a visual analogue scale (VAS) over a 72-hour period. The secondary outcomes will include adverse events associated with each medication, length of hospital stay, and the need for further interventions.

This study has the potential to provide important insights into the optimal management of pain in mild to moderate acute pancreatitis, which can ultimately improve patient outcomes and reduce the burden of this condition on the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of mild to moderate acute pancreatitis based on clinical and radiological criteria
* Moderate pain intensity (NRS score of 4-7)
* No history of allergy or intolerance to NSAIDs or opiates
* No history of opioid abuse or addiction

Exclusion Criteria:

* Severe acute pancreatitis requiring intensive care unit admission
* Pregnancy or lactation
* History of significant renal or hepatic dysfunction
* Use of non-steroidal anti-inflammatory drugs or opiates in the past 24 hours
* Known or suspected peptic ulcer disease
* Known or suspected gastrointestinal bleeding
* Participation in another clinical trial in the past 30 days
* Inability to provide informed consent
* Inability to communicate pain intensity using the numeric rating scale
* Allergy or intolerance to any of the study medications or their components.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity at 2 hours | 2 hours
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". The primary outcome of this study is pain intensity measured on the NRS at 2 hours after the intervention

SECONDARY OUTCOMES:
Pain intensity at 4, 6, 8, and 24 hours after the intervention | 4-24 hours
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable". Pain intensity will be measured at NRS scale at 4, 6, 8 and 24 hours after the intervention and recorded accordingly
time to pain relief | 0-24 hours
  How much time did it take for the pain to relieve completely. (In hours)
adverse events | 0-24 hours
  any adverse events with the drug intervention will be noted
patient satisfaction with pain management. | 1 day
  In this study, patient satisfaction with pain management will be assessed using a modified version of the Likert scale. Participants will be asked to rate their satisfaction with pain management on a scale from 1 to 5, where 1 is "very dissatisfied," 2 is "somewhat dissatisfied," 3 is "neither satisfied nor dissatisfied," 4 is "somewhat satisfied," and 5 is "very satisfied." This scale will be administered at 24 hours after the intervention.
  The satisfaction scale will also include an open-ended question to allow patients to provide any comments or suggestions regarding their pain management experience. These comments can provide valuable insights into the patient experience and help to inform future pain management practices.

CONTACTS AND LOCATIONS:
Overall Officials: Rehman Ullah Jan, Study Chair — Hayatabad Medical Complex
Locations (1):
- Hayatabad Medical Complex, Peshawar, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years
Access Criteria: The data will be shared on request by the institution